CLINICAL TRIAL: NCT04187079
Title: Immunopathologic Profiles of the Lung Micro- Environment Using Cryobiopsies and Identification of Blood Biomarkers in Patients With IPF
Brief Title: Immunopathologic Profiles and Blood Biomarkers in Patients With IPF
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Cryobiopsy in IPF
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Cryobiopsies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IPF: Patients diagnosed with idiopathic pulmonary fibrosis after multidisciplinary team discussion using medical history, HRCT pattern, laboratory findings, pulmonary function tests and cryobiopsy specimens.
- Other ILDs: Patients diagnosed with other interstitial diseases other than IPF after multidisciplinary team discussion using medical history, HRCT pattern, laboratory findings, pulmonary function tests and cryobiopsy specimens.

SUMMARY:
Examination of expression of PD-L1, PD-L2, Beta- catenin, B-cell follicles and Tenascin- C in patients with IPF compared with other interstitial lung diseases. Examination of anti HSP 70, p-ANCA, c-ANCA, CD4+/CD28- and CD8+/CD28- cells in patients with IPF compared with other interstitial lung diseases.

Compare the above mentioned findings with changes in pulmonary function tests, 6 minute walking test, exacerbation and mortality over a 2 year follow-up period.

DETAILED DESCRIPTION:
Examination of expression of PD-L1, PD-L2, Beta- catenin, B-cell follicles and Tenascin- C in cryobiopsies from the lungs inpatients with IPF compared with other interstitial lung diseases. Examination of anti HSP 70, p-ANCA, c-ANCA, CD4+/CD28- and CD8+/CD28- cells in blood samples in patients with IPF compared with other interstitial lung diseases.

Compare the above mentioned findings with changes in pulmonary function tests, 6 minute walking test, exacerbation and mortality over a 2 year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of having an ILD who are having cryobiopsies performed

Exclusion Criteria:

* BMI > 35
* DLCO < 35%
* FVC < 45%
* Pulmonary hypertension
* Cardiac or other severe comorbidity that will increase the risk of complications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of having an ILD who are having cryobiopsies performed to get a histological specimen for the diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
PD-L1 | At diagnosis
  Expression of PD-L1 in the epithelial cells in lungs

CONTACTS AND LOCATIONS:
Overall Officials: Venerino Poletti, Prof, Principal Investigator — Department of Respiratory Diaseses, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Respiratory Diseases and Allergy, Aarhus, Denmark